CLINICAL TRIAL: NCT04163666
Title: Effects of Mirror Therapy and Cognitive Therapeutic Exercise on Improvements to the Upper Member Functions of Stroke Patients: a Randomized Clinical Test Study Protocol
Brief Title: Effects of Mirror Therapy and Cognitive Therapeutic Exercise in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Burgos (Other)
Collaborators: Castilla-León Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBU-HUBU: MT-CTE
Record Dates: First submitted 2019-11-06; First posted 2019-11-15 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Stroke; Hemiparesis
Keywords: Stroke; Upper member; Neurorehabilitation; Mirror therapy; Therapeutic cognitive exercise; Perfetti
MeSH Terms: conditions — Stroke; Paresis | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mirror therapy group (Experimental): The mirror therapy group will receive a treatment based on this therapy, combined with task-oriented motor learning.
  Interventions: Behavioral: Mirror therapy
- Cognitive therapeutic exercise group (Experimental): The cognitive therapeutic exercise group will receive a treatment based on this therapy, combined with task-oriented motor learning.
  Interventions: Behavioral: Cognitive therapeutic exercise
- Control Group (No Intervention): No additional intervention with the participants of this group will be completed.

INTERVENTIONS:
Behavioral: Mirror therapy — The intervention will take place at the home of the participant for 6 weeks (30 days), during 60-minute sessions, 30 of which will be for mirror therapy, while the remaining 30 minutes will be for task-oriented motor learning
  Arms: Mirror therapy group
Behavioral: Cognitive therapeutic exercise — The intervention will take place at the home of the participant for 6 weeks (30 days), during 60-minute sessions, 30 of which will be for cognoscitive therapeutic exercise, while the remaining 30 minutes will be for task-oriented motor learning
  Arms: Cognitive therapeutic exercise group

SUMMARY:
This is a randomized clinical trial aimed at patients with a diagnosis of residual hemiparesis due to ischemic or hemorrhagic stroke. Its objective is to evaluate the effects of the mirror therapy and cognitive therapeutic exercise, both in combination with task-oriented motor learning, to achieve maximum functionality of the affected upper member,

DETAILED DESCRIPTION:
Objective: To assess the effect at 3 months of the of the mirror therapy and cognitive therapeutic exercise, both in combination with task-oriented motor learning, applied for 30 days in the functionality of the affected upper member, cognitive performance, emotional state, performance of daily living activities and quality of life in stroke patients.

Design and setting: A randomized clinical trial of three parallel groups.

Population: 152 patients with residual hemiparesis due to ischemic or hemorrhagic stroke will be included, selected by consecutive sampling at the Neurological Service and Stroke Unit of the University Hospital of Burgos (HUBU).

Measurements and intervention: Functionality of the affected upper member, cognitive performance, emotional state, performance of daily living activities and health-related quality of life will be evaluated. The intervention groups will receive a treatment based either on mirror therapy or on congnitive therapeutic exercise, both combined with task-oriented motor learning for 30 days. No additional intervention with the participants of the control group will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of residual hemiparesis due to ischemic or hemorrhagic stroke,
* Movements of the affected upper members classified between stages II and IV on the Brunnstrom Scale
* Score on the Montreal Cognitive Assessment (MOCA) scale equal to or over 26

Exclusion Criteria:

* Heminegligence
* Wernicke's aphasia
* Visual deficits (homonymous hemianopsia)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Functionality of the affected upper member. | 3 months
  Measurement by Fugl-Meyer Scale: Score between 0 (worst functionality) and 126 (best functionality)

SECONDARY OUTCOMES:
Spasticity of the upper member | 3 months
  Measurement by Ashworth Scale: Score between 0 (best situation) and 5 (worst situation)
Cognitive performance. | 3 months
  Measurement by Montreal Cognitive Assessment Scale: Score between 0 (worst cognitive situation ) and 30 (best cognitive situation)
Emotional state and quality of life. | 3 months
  Measurement by Post-Stroke Quality of Life Scale: Score between 30 (best state) and 155 (worst state)
Basic Daily Living Activities | 3 months
  Measurement by Functional Independence Measure - Functional Assessment Measure: Score between 30 (worst situation) and 210 (best situation)
Instrumental activities of daily living | 3 months
  Measurement by Lawton-Brody Index: Score between 0 (worst state) and 6 (best state)

CONTACTS AND LOCATIONS:
Overall Officials: Raul Soto-Camara, PhD, Principal Investigator — Burgos University; Jeronimo Gonzalez-Bernal, PhD, Principal Investigator — Burgos University
Locations (1):
- Universitary Hospital of Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Santos J, Soto-Camara R, Rodriguez-Fernandez P, Jimenez-Barrios M, Gonzalez-Bernal J, Collazo-Riobo C, Jahouh M, Bravo-Anguiano Y, Trejo-Gabriel-Galan JM. Effects of home-based mirror therapy and cognitive therapeutic exercise on the improvement of the upper extremity functions in patients with severe hemiparesis after a stroke: a protocol for a pilot randomised clinical trial. BMJ Open. 2020 Sep 25;10(9):e035768. doi: 10.1136/bmjopen-2019-035768. PMID 32978182